CLINICAL TRIAL: NCT01561235
Title: The Contribution of Gastrointestinal Appetite Hormones to Protein-induced
Brief Title: Protein Dose-repsonse Effect on GLP-1, PYY and Appetite in Male Subjects
Acronym: Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B243
Record Dates: First submitted 2012-03-13; First posted 2012-03-22 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Protein; Appetite; Satiety; Energi intake; Appetite regulating hormones; Dose-response
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Protein (Active Comparator): Energy content 3 or 4 MJ/meal, depending on the subject's individual daily energy requirements).
  Macronutrient content: Protein: 14 E%, Fat: 30 E% and carbohydrate: 56E%. The fibre content was similar in all three test meals. The test meals were served as pork/rice/mushroom pâtés, flavoured with thyme in order to blind differences in taste.
  Interventions: Other: Dose-reponse effect of protein on appetite and appetite-regulating hormones
- Medium-high protein (Experimental): Energy content 3 or 4 MJ/meal, depending on the subject's individual daily energy requirements).
  Macronutrient content: Protein: 25E%, Fat: 30 E% and carbohydrate: 45E%. The fibre content was similar in all three test meals. The test meals were served as pork/rice/mushroom pâtés, flavoured with thyme in order to blind differences in taste.
  Interventions: Other: Dose-reponse effect of protein on appetite and appetite-regulating hormones
- High Protein (Experimental): Energy content 3 or 4 MJ/meal, depending on the subject's individual daily energy requirements).
  Macronutrient content: Protein: 50 E%, Fat: 30 E% and carbohydrate: 20E%. The fibre content was similar in all three test meals. The test meals were served as pork/rice/mushroom pâtés, flavoured with thyme in order to blind differences in taste.
  Interventions: Other: Dose-reponse effect of protein on appetite and appetite-regulating hormones

INTERVENTIONS:
Other: Dose-reponse effect of protein on appetite and appetite-regulating hormones — 3-arm meal study for investigation of the mechanisms responsible for the satiating effects of protein in three isocaloric test meals with a protein content of 14, 25 or 50 E% protein. A possible 4-h dose-response effect of protein was investigated on a number of appetite-regulating hormones/peptides, together with changes in subjective appetite sensations and sensory desires were evaluated and ad libitum energy intake.

SUMMARY:
Dietary protein appears to be the most satiating and thermogenic macronutrient. However, how protein exerts its effect on appetite is not fully known. The effect have been suggested to be related to a higher oxidation rate of protein compared to carbohydrate and fat, and also to a greater thermogenic effect causing greater increase in core temperature. The involvement of peripheral appetite-regulating hormones has only been sparingly investigated.

The objective is to investigate the satiating effects of meals with varying content of meat-based protein and whether a dose-response effect can be found on appetite-regulating hormones and appetite ratings.

Design: 25 men will participate in the 3-way, randomized, double-blind, crossover study. The test meals is isocaloric with 30E% fat and increasing protein content at the expense of carbohydrate. Test meals are: normal protein content (NP, 14E% protein), medium-high protein content (MHP, 25E%), and high protein content(HP, 50E%). Four-hour subjective appetite ratings and blood samples will be assessed every half-hour. Subsequently, the subjects will served an ad libitum lunch.

DETAILED DESCRIPTION:
Dietary protein appears to be the most satiating and thermogenic macronutrient (7-11). However, how protein exerts its effect on appetite is not fully known. The effect have been suggested to be related to a higher oxidation rate of protein compared to carbohydrate and fat (12), and also to a greater thermogenic effect causing greater increase in core temperature (13). The involvement of peripheral appetite-regulating hormones has only been sparingly investigated (14). These studies have only included two preloads of different concentrations of protein. This is not an optimal design for investigating the protein dose-dependent effect as the threshold can have been reached in between the two concentrations. The effect of protein has mainly been investigated on glucagon-like peptide-1 (GLP-1), ghrelin, cholecystokinin (CCK), and generally after intake of protein below 35% of the energy content (35E%) (5;15-18). The relationship between these appetite-regulating hormones and appetite is still elusive due to contradicting results. Only one study has investigated the effect of protein preloads above 50E%. Bowen et al. (19) found that the high protein preloads could decrease the concentration of CCK and the rate of gastric emptying, which have been shown to enhance the satiating effect of food (20-22). Thus there is a need to examine the effect of protein on appetite-regulating hormones in a dose-response manner in order to detect whether there is an interaction between them and if they can be related to changes in subjective sensations of appetite and EI (14). This should be examined by comparing more than two isocaloric meals in which the protein content and one other macronutrient should vary whereas the third macronutrient should be kept fixed.

Thus, the objective of this study is to investigate the mechanisms responsible for the satiating effects of protein in three isocaloric test meals with a protein content of 14, 25 or 50 E% protein. A possible dose-response effect of protein is investigated on a number of appetite-regulating hormones/peptides, together with changes in ad libitum energy intake.

Design: 25 men will participate in the 3-way, randomized, double-blind, crossover study. The test meals is isocaloric with 30E% fat and increasing protein content at the expense of carbohydrate. Test meals are: normal protein content (NP, 14E% protein), medium-high protein content (MHP, 25E%), and high protein content(HP, 50E%). Four-hour subjective appetite ratings and blood samples will be assessed every half-hour. Subsequently, the subjects will served an ad libitum lunch.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* BMI: 18.5-40 kg/m2,
* Weight stable (within +/- 3 kg) two months prior to study inclusion,
* Non-smoking,
* Nonathletic,

Exclusion Criteria:

* BMI > 40 kg/m2,
* Change in smoking status,
* Daily or frequent use of medication,
* Suffering from metabolic diseases,
* Suffering from psychiatric diseases,
* Suffering from any other clinical condition, which would make the subject unfit to participate in the study,
* Blood pressure was above 150/90 mmHg,
* Hemoglobin < 8 mmol/l.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Acute 4-h changes from baseline in the postprandial concentration of GLP-1 | Measured on 3 seperate test days in a crossover design. Each test day was seperated by >4 weeks. On each test day GLP-1 was measured prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 240 minutes post intake
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 30, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples are analyzed for GLP-1. Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed.

SECONDARY OUTCOMES:
Acute 4-h changes from baseline in subjective appetite sensations using visual analogue scales | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day appetite sensations were measured prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 210, 240 minutes post intake.
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 30, 60, 90, 120, 150, 180, 210, 240 minutes post intake.
  Measured subjective appetite sensations of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to something sweet, salty, rich in fat, or meat/fish.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed.
Acute 4-h changes from baseline in the postprandial concentration of appetite regulating hormones/peptides | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day blood samples were collected prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 240 minutes post intake.
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 30, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples are or will be analyzed for glucagon, pancreatic polypeptide (PP), glucose-dependent insulinotropic polypeptide (GIP), peptid YY (PYY), ghrelin, CCK, amylin and apolipoprotein-IV.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed.
Acute 4-h changes from baseline in the postprandial concentration of glucose | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day blood samples were collected prior to the test meal (time 0) and 15, 30, 45, 60, 90, 120, 150, 180, 240 minutes post intake.
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 15, 30, 45, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples was analyzed for glucose.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed
Acute 4-h changes from baseline in the postprandial concentration of insulin | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day blood samples were collected prior to the test meal (time 0) and 15, 30, 45, 60, 90, 120, 150, 180, 240 minutes post intake.
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 15, 30, 45, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples was analyzed for insulin.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed
Acute 4-h changes from baseline in the postprandial concentrations of lipids | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day blood samples were collected prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 240 minutes post intake.
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 30, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples were analyzed for triglycerides, free fatty acids (FFA), total cholesterol, HDL-cholesterol.
  The concentration of low density lipoprotein (LDL) cholesterol will be estimated as described by Friedwald et al.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed
Acute 4-h changes from baseline in the body temperature | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day temperature was measured prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 210, 240 minutes post intake.
  Body temperature measurement were assessed at time 0, 30, 60, 90, 120, 150, 180, 210, 240 minutes post intake.
  Temperature was measured in the participants' ears (ThermoScan 6022, Braun GmbH, Kronberg, Germany).
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed
Rate of gastric emptying (4-h change from baseline in postprandial concentration of paracetamol) | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day blood samples were collected prior to the test meal (time 0) and 30, 60, 90, 120, 150, 180, 240 minutes post intake.
  The subjects drank 500 mg paracetamol desolved in 100 ml water together with the test meal.
  Blood samples were taken prior to the test meal (baseline). After initiation of the test meal blood samples were collected at time 30, 60, 90, 120, 150, 180, 240 minutes.
  Blood samples was analyzed for concentration of paracetamol.
  Data are planned to be statistically analyzed as repeated measurements in mixed linear models. Peak and time to peak will also be analyzed.
Rating of the organoleptic quality of the test meals | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day after completion of the test meal (approximately) time 15 minutes post intake) subjects rated the test meals
  After completion of the meal the subjects rated the organoleptic quality of the meal by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability of the meal.
Rating of the organoleptic quality of the ad libitum meal | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day after completion of the ad libitum meal subjects rated the meal
  After completion of the meal the subjects rated the organoleptic quality of the ad libitum meal by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability of the meal.
Subjective appetite sensations (visual analogue scales) after ad libitum meal | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. On each test day after completion of the ad libitum meal subjects rated their subjective sensation of appetite (approximately 4.5-h post intake of the test meal)
  After completion of the meal the subjects rated the subjective appetite sensations by visual analogue scales (VAS) in regard to sensation of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to eat something sweet, salty, rich in fat, or meat/fish.
ad libitum energy intake (EI) | Measured on 3 seperate test days in a crossover design. Each test seperated by >4 weeks. EI was measured 240 min after intake of the test meal
  240 min after each test meal an ad libitum meal was served, and the total energy intake was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Dr Med, Principal Investigator — Depertment of Human Nutrition, University of Copenhagen, Denmark
Locations (1):
- Department of human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Belza A, Ritz C, Sorensen MQ, Holst JJ, Rehfeld JF, Astrup A. Contribution of gastroenteropancreatic appetite hormones to protein-induced satiety. Am J Clin Nutr. 2013 May;97(5):980-9. doi: 10.3945/ajcn.112.047563. Epub 2013 Mar 6. PMID 23466396